CLINICAL TRIAL: NCT02298062
Title: Infliximab for Kawasaki Disease Patients Resistant to Intravenous Immunoglobulin : a Multicentre, Prospective, Randomised Trial
Brief Title: Infliximab for Kawasaki Disease Patients Resistant to IVIG : a Multicentre, Prospective, Randomised Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Shanghai Children's Medical Center (Other); Shanghai 10th People's Hospital (Other); Shanghai 8th People's Hospital (Other); Shanghai Xuhui Distrct Center Hospital (Unknown)
Responsible Party: Principal Investigator, Fang liu, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-LF
Record Dates: First submitted 2014-09-23; First posted 2014-11-21 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2014-12

CONDITIONS: Kawasaki Disease
Keywords: Kawasaki disease coronary artery lesion, IVIG- resistant, Infliximab
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Infliximab; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infliximab (Experimental): For one group of patients with resistance to intravenous immunoglobulin in Kawasaki disease , we will give them infliximab (5mg/kg) once.
  Interventions: Drug: Infliximab
- IVIG (Active Comparator): For the other group of patients with resistance to intravenous immunoglobulin in Kawasaki disease , we will give them IVIG (2g/kg) once.
  Interventions: Drug: IVIG

INTERVENTIONS:
Drug: Infliximab — The treatment-resistant children will be randomly assigned to either the infliximab or IVIG group in a 1:1 ratio and receive either infliximab (5 mg/kg at 1 mg/mL intravenously over 2 h) or IVIG (2g/kg). The primary outcome measure is change in absolute cell counts, concentrations of C-reactive protein, alanine transaminase,IL-1,IL-6,TNF-a,STNFR-I,STNFR-2; number of fever days (24 h period with a temperature of at least 38•0°C) from enrolment; duration and cost of hospital stay.The secondary 0utcome Measure is the incidence of coronary artery abnormalities
  Arms: Infliximab
Drug: IVIG — The treatment-resistant children will be randomly assigned to either the infliximab or IVIG group in a 1:1 ratio and receive either infliximab (5 mg/kg at 1 mg/mL intravenously over 2 h) or IVIG (2g/kg). The primary outcome measure is change in absolute cell counts, concentrations of C-reactive protein, alanine transaminase,IL-1,IL-6,TNF-a,STNFR-I,STNFR-2; number of fever days (24 h period with a temperature of at least 38•0°C) from enrolment; duration and cost of hospital stay.The secondary 0utcome Measure is the incidence of coronary artery abnormalities
  Arms: IVIG

SUMMARY:
The objective of this study is to investigate the effect of infliximab to the children who don't respond to the first dose of intravenous immunoglobulin (IVIG) (2g/kg) in Kawasaki disease.

DETAILED DESCRIPTION:
Kawasaki disease(KD), the most common cause of acquired heart disease in developed countries, is a self-limited vasculitis that is treated with high doses of intravenous immunoglobulin. Resistance to intravenous immunoglobulin in Kawasaki disease which is defined as a temperature of 38.0°C or higher at 36 hours to 7 days after completion of the infusion of intravenous immunoglobulin increases the risk of coronary artery lesions. We will conduct a multicenter, randomized, prospective trial to determine whether the use of infliximab to the children who don't respond to the first dose of IVIG(2g/kg) reduces the risk of coronary artery diseases. The IVIG-resistant children will be randomly assigned to either the infliximab or IVIG group in a 1:1 ratio and receive either infliximab (5 mg/kg at 1 mg/mL intravenously over 2 h) or IVIG (2g/kg). The level of leukocyte (WBC)counts, C-reactive protein, alanine transaminase,interleukin- 1( IL-1), interleukin- 6(IL-6), tumor necrosis factor-a(TNF-a), soluble tumor necrosis factor receptor-1(STNFR-I), soluble tumor necrosis factor receptor-2(STNFR-2), the fever days,and the cost of hospital stay will be analyzed between these two groups.The final outcome is the incidence of coronary artery lesions.

ELIGIBILITY:
Inclusion Criteria:

* (1)Individual patient's medical file data confirmed the diagnosis of KD using the 5th revised edition of diagnostic criteria for KD, issued by the Japan Kawasaki Disease Research Committee at the 7th International Kawasaki Disease Symposium in 2002.(2) Resistance to intravenous immunoglobulin in Kawasaki disease is defined as a temperature of 38.0°C or higher at 36 hours to 7 days after completion of the routine primary treatment .(3) the patients aged from 2 months to 12 years old. (4) All included patients required to sign an informed consent form

Exclusion Criteria:

. Exclusion criteria: (1) The patients with severe infections; (2) The patients with a history of tuberculosis or recent close contact with tuberculosis; (3) The patient vaccinated with live vaccine in 6 months; (4)The patients with the application of hormone or other immunosuppressive agents; (5) The patients didn"t want to signed informed consent.

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
change in concentrations of cytokines | 2 years
  we will obtain laboratory data including concentrations of C-reactive protein, alanine transaminase,IL-1,IL-6,TNF-a,STNFR-I,STNFR-2 at baseline, 72 h after completion of the intravenous immunoglobulin infusion, and at week 2 and week 4 after randomisation.

SECONDARY OUTCOMES:
incidence of coronary artery lesions(CAL) | 2 years
  Echocardiography is performed in the acute phase ,early and late recovery of Kawasaki disease

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China